CLINICAL TRIAL: NCT03803917
Title: Treatment of Perianal Fistulas in Crohn's Disease With Injection of Freshly Harvested Autologous Adipose Tissue
Brief Title: Adipose Tissue in Crohn´s Disease Fistulas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lilli Lundby (Other)
Responsible Party: Sponsor-Investigator, Lilli Lundby, Principal investigator, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT_ Fistula_observational
Record Dates: First submitted 2019-01-08; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Crohn Disease; Perianal Fistula; Tissue Transplantation
MeSH Terms: conditions — Crohn Disease | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Other): Injection with freshly collected autologous adipose tissue
  Interventions: Procedure: Injection with freshly collected autologous adipose tissue

INTERVENTIONS:
Procedure: Injection with freshly collected autologous adipose tissue

SUMMARY:
Present study investigated the efficacy of injection of freshly collected autologous adipose tissue into perianal fistulas in patients with Crohn's disease. Adipose tissue collected by liposuction was injected into the perianal fistulas. Primary objective was complete clinical healing six months after treatment. Secondary objectives were reduced or ceased fistula secretion and complications to the treatment.

DETAILED DESCRIPTION:
Investigators prospectively registered symptoms, complications and results of treatment in 21 patients with Crohn´s Disease who underwent treatment with freshly harvested autologous adipose tissue for perianal fistulas between March 2015 and June 2018. Inclusion criteria consisted of the following: the presence of complex CD fistulas refractory to standard surgical intervention, including long-term seton and regular curettage, and/or medical treatment. Pelvic magnetic resonance imaging (MRI) was performed to describe the location and extent of the fistula. Clinical examinations of the patients were performed at intervals of six weeks, three months and six months following adipose tissue injection. Primary endpoint was complete fistula healing at clinical examination six months after the last injection. A fistula was considered completely clinically healed: (i) if the patient had no symptoms of discharge; (ii) if there was no visible external fistula opening in the perineum; and (iii) if no internal opening could be palpated with rectal digital examination. Secondary endpoints included either reduced or ceased fistula secretion. If clinical healing of the fistula was not obtained six weeks after the first treatment, patients were offered a second adipose injection within two weeks. A third injection was offered to patients who did not have complete healing within six weeks of the first two injections.Pelvic MRI was repeated in all patients with transsphincteric and intersphincteric fistulas who, upon clinical examination, demonstrated complete healing at 6 months after the last injection.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Crohn´s Disease
* presence of complex Crohn´s Disease fistulas
* fistulas refractory to standard surgical intervention, including long-term seton and regular curettage, and/or medical treatment.

Exclusion Criteria:

- Fistulas developed following proctectomy were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-03-01; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical healing | 6 months after last injection
  A fistula was considered completely clinically healed: (i) if the patient had no symptoms of discharge; (ii) if there was no visible external fistula opening in the perineum; and (iii) if no internal opening could be palpated with rectal digital examination

SECONDARY OUTCOMES:
Ceased or reduced fistula secretion | 6 months after last injection
  Reported by the individual patient
Complications to the treatment | 6 months after last injection
  Reported by the individual patient and findings by clinical examination

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dige A, Hougaard HT, Agnholt J, Pedersen BG, Tencerova M, Kassem M, Krogh K, Lundby L. Efficacy of Injection of Freshly Collected Autologous Adipose Tissue Into Perianal Fistulas in Patients With Crohn's Disease. Gastroenterology. 2019 Jun;156(8):2208-2216.e1. doi: 10.1053/j.gastro.2019.02.005. Epub 2019 Feb 14. PMID 30772343